CLINICAL TRIAL: NCT01901991
Title: A Randomized Study of Localization of Nonpalpable Breast Lesions - RSL vs WGL
Brief Title: Localization of Nonpalpable Breast Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Linnea Langhans, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R72-A4701-13-S9
Record Dates: First submitted 2013-07-14; First posted 2013-07-17 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2016-09

CONDITIONS: Breast Cancer; Carcinoma in Situ
Keywords: Nonpalpable breast lesions; Breast Cancer and carcinoma in situ; Radioactive seed localization; Wire-guided localization; Randomized study
MeSH Terms: conditions — Breast Neoplasms; Carcinoma in Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radioactive seed localization (RSL) (Experimental): Patients are randomised for preoperative lesion localization with either radioactive seed localization (RSL) or wire-guided localization (WGL).
  In this arm 205 patients will have RSL performed. The radioactive seed is introduced through a gauge needle using standard ultrasound guidance. Once guided to the nonpalpable breast lesion, the seed is deployed into the breast tissue by advancing a stilette in the needle. The exact location is confirmed by mammography. The nonpalpable lesion is located during the operation with a handheld gamma probe, identical to the one used for the sentinel node procedure. The surgical specimen is orientated and examined at the Department of Radiology and Pathology in accordance with the existing guidelines of WGL.
  Interventions: Procedure: Radioactive seed localization (RSL)
- Wire-guided localization (WGL) (Active Comparator): Patients are randomised for preoperative lesion localization with either radioactive seed localization (RSL) or wire-guided localization (WGL).
  In this arm 205 patients will have WGL performed. Guided by ultrasound or mammography a flexible wire is introduced into the breast by the radiologist just before the operation. The tip of the wire must mark the nonpalpable lesion, and correct localization is verified by mammography. The surgeon uses the wire and mammography as a guide during the operation. The surgical specimen is orientated and examined at the Department of Radiology and Pathology in accordance with the existing guidelines of WGL.
  Interventions: Procedure: Wire-guided localization (WGL)

INTERVENTIONS:
Procedure: Radioactive seed localization (RSL) — Localization of nonpalpable breast lesions with Radioactive seed localization
  Arms: Radioactive seed localization (RSL)
Procedure: Wire-guided localization (WGL) — Localization of nonpalpable breast lesions with Wire-guided localization
  Arms: Wire-guided localization (WGL)

SUMMARY:
Each year the Danish mammography-screening programme identifies a large number of patients with small non-palpable breast cancers or precancerous lesions. The majority of these patients are suitable for breast conserving surgery (BCS). The object of BCS is to remove the suspicious lesion completely without removing excess healthy breast tissue. To obtain this accurate lesion localization is essential.

Until today the standard procedure in Denmark has been wire guided localization (WGL). Although the method has been utilized for a number of years it has several disadvantages. Often inaccurate lesion localization leads to incomplete lesion removal (positive margin) and subsequently reoperation. It can postpone the additional systemic treatment, offered after the operation. Other disadvantages are poor cosmetic outcome and inconvenient planning for the patient and the departments involved. The wire needs to be placed on the day of the operation, which decreases the flexibility of the procedure.

The purpose of this study is to test a new method named radioactive seed localization (RSL). The method uses a small titanium seed containing radioactive iodine. It will be placed in the centre of the lesion, and during the operation, the surgeon can locate it with a handheld gamma probe. The seed can be placed a few days in advance, which means a more flexible course of treatment. The method seems promising with regards to reoperation rates, but it needs further testing.

Hypothesis:

RSL is a more accurate method, for localization of nonpalpable breast lesions, than WGL. Using RSL obtains, to a great extent, adequate negative margins, resulting in a reduced number of re-operations.

The study will be performed as a randomised clinical trial, where the two methods will be compared to each other. The trial will be performed at the department of breast surgery at Rigshospitalet and include patients with nonpalpable breast lesions. Besides reoperation rates, duration of the surgical procedure and the amount of removed breast tissue will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nonpalpable breast lesions, carcinoma in situ or invasive carcinoma, where preoperative lesion localization is necessary.
* All age groups, minimum 18 years

Exclusion criteria:

* Patients with benign nonpalpable breast lesions.
* Patients who are unable to comprehend the information.
* Patients who are pregnant, breastfeeding or have children < 3 years.
* Patients who have lesions, which requires more than two wires or seeds for localization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Re-operation rate due to positive microscopic margins detected at the final pathological evaluation. | Re-operation within 3 months after the initial breast conserving surgery.

SECONDARY OUTCOMES:
Amount of excised breast tissue in relation to tumour size. | 3 months.

OTHER OUTCOMES:
Duration of the surgical procedure. | 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Kroman, Professor, Study Chair — Rigshospitalet (Copenhagen University Hospital), Department of Breast Surgery
Locations (1):
- Rigshospitalet (Copenhagen University Hospital), Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented in a international peer review article.

REFERENCES:
- [Result] Langhans L, Tvedskov TF, Klausen TL, Jensen MB, Talman ML, Vejborg I, Benian C, Roslind A, Hermansen J, Oturai PS, Bentzon N, Kroman N. Radioactive Seed Localization or Wire-guided Localization of Nonpalpable Invasive and In Situ Breast Cancer: A Randomized, Multicenter, Open-label Trial. Ann Surg. 2017 Jul;266(1):29-35. doi: 10.1097/SLA.0000000000002101. PMID 28257326